CLINICAL TRIAL: NCT02960048
Title: Clinical Evaluation of Stabilizing Splint (Michigan-type Occlusal Splint) Versus Anterior Repositioning Splint in Patients With Temporomandibular Joint Anterior Disc Displacement With Reduction . ( Randomized Controlled Clinical Study)
Brief Title: Clinical Evaluation of Stabilizing Splint (Michigan-type Occlusal Splint) Versus Anterior Repositioning Splint .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Moataz Nasr, Oral and maxillofacial surgery resident in Sahel Teaching hospital, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CairoARS-SRS
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: TMJ Disc Disorder
Keywords: Anterior disc displacement; TMD therapy; internal derangement; occlusal splint; anterior repositioning splint

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior repositioning splint (Active Comparator): A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch .
  Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient is instructed to protrude the mandible slightly and to open and close the mouth In this position.
  Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop .
  Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe.
  Interventions: Device: Anterior repositioning splint
- Stabilizing splint (Experimental): A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch .
  Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient should be instructed to close in Centric relation . Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop .
  Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe. All areas, except labial to the mandibular canines, are flattened to the contact marks. This area will create the eccentric guidance.
  Interventions: Device: Stabilizing splint

INTERVENTIONS:
Device: Stabilizing splint — A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch .
  Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient should be instructed to close in Centric relation . Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop .
  Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe. All areas, except labial to the mandibular canines, are flattened to the contact marks. This area will create the eccentric guidance.
  Other Names: Michigan-type occlusal splint
  Arms: Stabilizing splint
Device: Anterior repositioning splint — A 2-mm-thick, hard, clear sheet of resin will be adapted to the maxillary arch .
  Small amount of self-curing acrylic will be added to the anterior portion of the appliance as a stop for the lower incisor. The area of this stop is approximately 4 to 6 mm. The patient is instructed to protrude the mandible slightly and to open and close the mouth In this position.
  Self-curing acrylic will be added to the occluding surface of the appliance. All occluding areas, except the contact on the anterior stop .
  Excess acrylic surrounding the centric contacts is removed with a hard rubber wheel on a lathe.
  Other Names: ARS
  Arms: Anterior repositioning splint

SUMMARY:
To evaluate the effectiveness of Michigan-type occlusal splint and anterior repositioning splint in patients with temporomandibular joint anterior disc displacement with reduction.

DETAILED DESCRIPTION:
To evaluate the effectiveness of Michigan-type occlusal splint and anterior repositioning splint in patients with temporomandibular joint anterior disc displacement with reduction.

PICO:

Population (P): Patients with symptomatic anterior disc displacement with reduction.

Intervention (I): Michigan splint. Comparator (C): Anterior repositioning splint (ARS) .

Outcome(O):

Primary outcome: Patients' subjective pain experience. Each patient will be asked to rate his or her current and worst pain intensity on numerical rating scale (NRS) of 0-10 with zero being no pain and ten corresponds to the worst pain that the patient ever had.

Secondary outcome:

1. Maximum mouth opening (MMO). Assessment of MMO will be performed by measuring the distance in mm between the incisal edges of the upper and lower central incisors using a ruler.
2. lateral excursion . Assessment of lateral excursion will be performed by measuring the distance in mm between midline of upper and lower jaws
3. protrusion. distance in mm from the incisal edge of the maxillary central incisor to the incisor edge of the mandibular incisor will measured in the maximum protruded position.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient from 15 to 50 years old.
2. Report of pain in preauricular region worsened by functional activities, such as chewing and talking.
3. Presence of disc displacement with reduction and joint clicking
4. positive diagnosis of unilateral or bilateral anterior disc displacement with reduction by means of magnetic resonance imaging (MRI).

Exclusion Criteria:

1. . .
2. History of TMJ surgery.
3. Individuals with osteoarthritis.
4. Individuals under TMD management.
5. Individuals wearing full or partial dentures.
6. Individuals with major psychological disorders.
7. Nonreducing dislocations of the articular disc
8. Consequences of condyle fractures and/or fracture of another maxillofacial zone.
9. Articular pathologies of systemic nature (e.g., rheumatoid arthritis, arthrosis, psoriasis arthritis).
10. Individuals with a recent history of trauma in the face and/or neck area. Individuals with systemic diseases that can affect TMJ

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Patients' subjective pain experience. | 3 months
  Each patient will be asked to rate his or her current and worst pain intensity on numerical rating scale (NRS) of 0-10 with zero being no pain and ten corresponds to the worst pain that the patient ever had.

SECONDARY OUTCOMES:
Maximum mouth opening. | 3 months
  measuring the distance between the incisal edges of the upper and lower central incisors using a ruler.Unit:mm
Lateral excursion. | 3 months
  measuring the distance between midline of upper and lower jaws . Unit: mm
Protrusion. | 3 months
  The distance in mm from the incisal edge of the maxillary central incisor to the incisor edge of the mandibular incisor will measured in the maximum protruded position.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Galal, MD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebrahim S, Montoya L, Busse JW, Carrasco-Labra A, Guyatt GH; Medically Unexplained Syndromes Research Group. The effectiveness of splint therapy in patients with temporomandibular disorders: a systematic review and meta-analysis. J Am Dent Assoc. 2012 Aug;143(8):847-57. doi: 10.14219/jada.archive.2012.0289. PMID 22855899
- [Background] Huang IY, Wu JH, Kao YH, Chen CM, Chen CM, Yang YH. Splint therapy for disc displacement with reduction of the temporomandibular joint. part I: modified mandibular splint therapy. Kaohsiung J Med Sci. 2011 Aug;27(8):323-9. doi: 10.1016/j.kjms.2011.03.006. Epub 2011 May 10. PMID 21802643
- [Background] Lundh H, Westesson PL, Kopp S, Tillstrom B. Anterior repositioning splint in the treatment of temporomandibular joints with reciprocal clicking: comparison with a flat occlusal splint and an untreated control group. Oral Surg Oral Med Oral Pathol. 1985 Aug;60(2):131-6. doi: 10.1016/0030-4220(85)90280-4. PMID 3862019
- [Background] Badel T, Marotti M, Kern J, Laskarin M. A quantitative analysis of splint therapy of displaced temporomandibular joint disc. Ann Anat. 2009 Jun;191(3):280-7. doi: 10.1016/j.aanat.2008.12.004. Epub 2009 Feb 12. PMID 19282162
- [Background] Conti PC, Correa AS, Lauris JR, Stuginski-Barbosa J. Management of painful temporomandibular joint clicking with different intraoral devices and counseling: a controlled study. J Appl Oral Sci. 2015 Oct;23(5):529-35. doi: 10.1590/1678-775720140438. Epub 2015 Jul 21. PMID 26200526
- [Background] Conti PC, de Azevedo LR, de Souza NV, Ferreira FV. Pain measurement in TMD patients: evaluation of precision and sensitivity of different scales. J Oral Rehabil. 2001 Jun;28(6):534-9. doi: 10.1046/j.1365-2842.2001.00727.x. PMID 11422679
- [Background] Khare N, Patil SB, Kale SM, Sumeet J, Sonali I, Sumeet B. Normal mouth opening in an adult Indian population. J Maxillofac Oral Surg. 2012 Sep;11(3):309-13. doi: 10.1007/s12663-012-0334-1. Epub 2012 Feb 19. PMID 23997482
- [Background] Sharmila devi Devaraj 1 and 2, "Internal Derangement of Temporomandibular Joint - A Review\n," IOSR J. Dent. Med. Sci., vol. 13, no. 3, pp. 66-73, 2014.
- [Background] T. Badel, V. Lajnert, and D. Zadravec, "Michigan splint and treatment of temporomandibular joint Michiganska udlaga i liječenje temporomandibularnog zgloba," vol. 49, no. 2, pp. 112-120, 2013.
- See also: Related Info — http://doi.org/10.1007/s12663-012-0334-1
- See also: Related Info — http://doi.org/10.1590/1678-775720140438